CLINICAL TRIAL: NCT02165787
Title: Investigation of Gait Parameters in Health and Neurological Disease Under Varying Locomotor Conditions
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2014-0004/PB_2016-00386
Record Dates: First submitted 2014-05-23; First posted 2014-06-17 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Gait Analysis in Neurological Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- patients
- healthy control subjects

SUMMARY:
In the cross-sectional component of this study, our overall objective is to gather a large pool of data from which we can generate gait "profiles". These profiles will consist of a constellation of gait (+/- electrophysiological) parameters associated with a particular neurological diagnosis or specific lesion(s) in neuroanatomical systems. Once developed, these profiles can be compared for differences and similarities; allowing insights into the specificity of the effect on gait of a given diagnosis or lesion in the case of the former and redundancy of neuroanatomical systems in that of the latter. A longitudinal component of the study will look at the evolution of gait parameters over time in a group of patients with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* age 18 - 80
* written, informed consent
* one of the following established diagnoses: unilateral stroke affecting motor system, Parkinson syndrome, cerebellar disease, vestibular dysfunction, spinal cord injury, multiple sclerosis
* Brain and whole spine T1, T2 & FLAIR magnetic resonance imaging performed within the last four months and available for study purposes or no contraindications to performing these scans

Healthy subjects:

* age 18 - 80
* written informed consent

Exclusion Criteria:

Patients:

* Colour-blindness
* Known to be pregnant or breastfeeding
* Body mass index (weight in kg/height in metres squared) >40 Unable to walk 50m within 6 minutes (with or without walking aids) Inability to undertake any component of the trial protocol
* Terminal diagnosis with life expectancy less than six months
* Cognitive disturbance defined as MMSE < 25 Clinically significant comorbidities such as severe cardiovascular, pulmonary or malignant disease

Healthy subjects:

* Colour-blindness
* Known to be pregnant or breastfeeding
* Body mass index (weight in kg/height in metres squared) >40 Unable to walk 50m within 6 minutes
* Reliance on walking aids / prostheses for mobilisation
* Significant neurological or orthopaedic diagnosis with potential impact on gait // Previous operations on the lower limbs or spine with potential impact on gait Inability to undertake any component of the trial protocol Clinically significant conditions such as severe cardiovascular, pulmonary or malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-80 with spinal cord injury, hemispheric stroke, multiple sclerosis, Parkinson disease, vestibular disease, cerebellar disease. Healthy control subjects aged 18-80.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2014-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Change of gait parameter after injury to CNS | Timepoint 0 plus timepoint 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Killeen T, Easthope CS, Filli L, Linnebank M, Curt A, Bolliger M, Zorner B. Modulating Arm Swing Symmetry with Cognitive Load: A Window on Rhythmic Spinal Locomotor Networks in Humans? J Neurotrauma. 2017 May 15;34(10):1897-1902. doi: 10.1089/neu.2016.4554. Epub 2016 Oct 12. PMID 27574966
- [Background] Killeen T, Easthope CS, Filli L, Lorincz L, Schrafl-Altermatt M, Brugger P, Linnebank M, Curt A, Zorner B, Bolliger M. Increasing cognitive load attenuates right arm swing in healthy human walking. R Soc Open Sci. 2017 Jan 25;4(1):160993. doi: 10.1098/rsos.160993. eCollection 2017 Jan. PMID 28280596
- [Background] Filli L, Meyer C, Killeen T, Lorincz L, Gopfert B, Linnebank M, von Tscharner V, Curt A, Bolliger M, Zorner B. Probing Corticospinal Control During Different Locomotor Tasks Using Detailed Time-Frequency Analysis of Electromyograms. Front Neurol. 2019 Jan 29;10:17. doi: 10.3389/fneur.2019.00017. eCollection 2019. PMID 30761064
- [Background] Killeen T, Easthope CS, Demko L, Filli L, Lorincz L, Linnebank M, Curt A, Zorner B, Bolliger M. Minimum toe clearance: probing the neural control of locomotion. Sci Rep. 2017 May 15;7(1):1922. doi: 10.1038/s41598-017-02189-y. PMID 28507300